CLINICAL TRIAL: NCT03118011
Title: Tobacco Habits and the Ability to Quit Smoking Among Patients With Substance Use Disorders
Brief Title: Substance Use Disorders and Tobacco Habits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Katarina Danielsson, Medical Doctor, Doctor of Philosphy (Faculty of Medicine), Uppsala University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/048
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Substance Use Disorders
Keywords: Tobacco use, withdrawal symptoms
MeSH Terms: conditions — Substance-Related Disorders; Tobacco Use; Substance Withdrawal Syndrome | interventions — Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No smoking (Active Comparator): The ward where the patients can not go out to smoke
  Interventions: Other: No smoking
- Smoking (Placebo Comparator): The ward where the patients can go out to smoke.
  Interventions: Other: Smoking

INTERVENTIONS:
Other: No smoking — No smoking
  Arms: No smoking
Other: Smoking — Ability to go out to smoke
  Arms: Smoking

SUMMARY:
In the department for substance use disorders at Uppsala University Hospital there are two wards. One that is locked, where the patients that are emitted can not go out to smoke and another ward where there is a possibility to go out and smoke during the day.

The smoking habits on those two floors will be compared and how they feel about smoking will be evaluated when they are admitted to the ward, at discharge, after 1 mont and after 6 months.

DETAILED DESCRIPTION:
In the department for substance use disorders at Uppsala University Hospital there are two wards. One that is locked, where the patients that are emitted can not go out to smoke and another ward where there is a possibility to go out and smoke during the day.

The smoking habits on those two wards will be compared and how they feel about smoking will be evaluated when they are admitted to the ward, at discharge, after 1 mont and after 6 months.

The questionnaires that will be used for evaluation are:

Fagerstöms test for nicotine dependence, Alcohol Use Disorders Identification Test and Drug Use Disorders Identification Test and the symptoms of Tobacco withdrawal mentioned in DSM-V.

Parameters that will be measured are: pulse, bloodpressure, peak expiratory flow, wight and height.

There will also be some questions about their smoking and snuff habits, if they have tried to quite smoking Before and how they were affected by the stop.

ELIGIBILITY:
Inclusion Criteria: Substance use disorder -

Exclusion Criteria: Disorganization, psychosis and if you can not speak Swedish.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Less smoking | From baseline to 1 month
  Number of cigarettes /day
Less smoking | From baseline to 6 month
  Number of cigarettes /day

SECONDARY OUTCOMES:
withdrawal symptoms | From baseline to emitted from the ward aproximately 1 week
  Blood pressure, Worry, nausea e.t.c.
withdrawal symptoms | From baseline to 1 month
  Blood pressure, Worry, nausea e.t.c.
withdrawal symptoms | From baseline to 6 month
  Blood pressure, Worry, nausea e.t.c.
Thought about not smoking any more | From baseline to emitted from the ward aproximately 1 week
  Questions
Thought about not smoking any more | From baseline to 1 month
  Questions
Thought about not smoking any more | From baseline to 6 month
  Questions
PEF | From baseline to emitted from the ward aproximately 1 week
  Improved expiratory flow
PEF | From baseline too 1 month
  Improved expiratory flow
PEF | From baseline to 6 month
  Improved expiratory flow
Weight | From baseline to emitted from the ward aproximately 1 week
  Changes in weight
Weight | From baseline to 1 month
  Changes in weight
Weight | From baseline to 6 month
  Changes in weight

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Danielsson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No